CLINICAL TRIAL: NCT01916304
Title: A Multicentre, Open-label Switch Study to Investigate the Necessity of Dose Adjustment After Switching From L-Thyroxine Christiaens® to the New Levothyroxine Sodium Test Formulation in (Near) Total Thyroidectomised Patients.
Brief Title: Study of Dose Adjustment From Levothyroxine to a New Levothyroxine Sodium Test Formulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LE-9999-401-BE; 2012-005732-28 (EudraCT Number); U1111-1145-3526 (Registry Identifier: UTN (WHO))
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-06

CONDITIONS: Hypothyroidism
Keywords: Drug Therapy
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levothyroxine sodium new formulation (Experimental): Levothyroxine (25-225 μg), tablets, orally, once daily for up to 12 to 20 weeks. Dose administered depends on the thyroid stimulating hormone level.
  Interventions: Drug: Levothyroxine sodium new formulation

INTERVENTIONS:
Drug: Levothyroxine sodium new formulation — Levothyroxine tablets

SUMMARY:
The purpose of this study is to investigate the effect of switching participants taking levothyroxine to a new sodium formulation.

DETAILED DESCRIPTION:
The drug being tested in this study is a new sodium formulation of levothyroxine. Levothyroxine (L-Thyroxine Christiaens®) is used in the treatment of hypothyroidism. This study will investigate the effect of switching subjects taking levothyroxine to a new levothyroxine sodium formulation.

The results of this study will be used to provide instructions to general practitioners and endocrinologists assisting patients on levothyroxine hormone substitution in performing the switch to the new formulation.

The study will enroll approximately 90 patients. Patients receiving the same daily dose of L-Thyroxine Christiaens® during the past 6 weeks and with serum thyroid stimulating hormone (TSH) levels between 0.4-2.5 mU/L will be switched to the equivalent daily dose of the new formulation of levothyroxine. After the switch, patients will be followed up after 2 (± 2 weeks) and 4 months (± 4 weeks).

All participants will be asked to take a daily dose at the same time each day throughout the study.

This study will be conducted in Belgium. Participants will make 3 to 4 visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. (Near) total thyroidectomised patients.
2. Aged 18 years and older.
3. Stabilised on the same daily dose of L-Thyroxine Christiaens® during the last 6 weeks before inclusion in the study.
4. Written informed consent given.
5. Able and willing to comply with protocol requirements and to complete the study.

Exclusion Criteria:

1. History of Graves' disease or positive TSH-receptor antibodies.
2. History of thyroid cancer requiring TSH suppression.
3. Medical procedures or treatments planned that could influence the thyroid hormone state of the patients during this trial.
4. Use of levothyroxine containing medicines provided by other brands to treat hypothyroidism.
5. Pregnant or planning pregnancy. Female patients of childbearing potential need to apply highly effective methods of birth control.
6. Participation in another trial in the past 6 weeks.
7. Exclusion criteria during the study are the occurrence of any serious adverse reaction, any laboratory or clinically relevant change in patient status, any change in smoking status, use of drugs non-authorized by the physician (to avoid relevant drug interactions) and lack of patient compliance with the study drug. (OR events not considered as exclusion criteria but to be documented in the case report form, as a possible explanation for change in lab parameters and/or dose switch).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Takeda
Locations (1):
- Leuven, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in Belgium from 02 July 2013 (first patient screened) to 23 June 2014.
Pre-assignment Details: Participants with a diagnosis of Primary Hypothyroidism were switched from treatment with L-Thyroxine Christiaens® to treatment with new levothyroxine sodium 25-225 μg.
Period: Overall Study
Arm/Group | Levothyroxine Sodium New Formulation
Started | 101
Safety Set | 101
Intent-to-Treat Set | 84
Completed | 84
Not Completed | 17
Not completed — Screening failure | 17

BASELINE CHARACTERISTICS:
Arm/Group | Levothyroxine Sodium New Formulation
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (12.17)
Age, Customized [Number; unit: participants]
  <65 years | 78
  ≥ 65 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 29
Region of Enrollment [Number; unit: participants]
  Belgium | 101
Weight [Mean (Standard Deviation); unit: kg] — Weight data is available for 100 participants.
  kg | 76.9 (18.05)
Height [Mean (Standard Deviation); unit: cm] — Height data was available for 96 participants.
  cm | 168.4 (8.57)
Investigator Reported Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Investigator reported BMI data was available for 93 participants.
  kg/m^2 | 27.2 (5.98)
Calculated BMI [Mean (Standard Deviation); unit: kg/m^2] — Calculated BMI data was available for 96 participants.
  kg/m^2 | 27.1 (6.00)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Do Not Need a Change of Dose
Description: Dose change was determined by physician according to their clinical judgement.
Time Frame: 2 months (± 2 weeks) after switch to sodium formulation.
Population: Participants from the intent-to-treat population, with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Levothyroxine Sodium New Formulation
Number analyzed (Participants) | 82
percentage of participants | 32.9 [23.7 to 43.7]

2. Secondary Outcome: Magnitude of the Change in Daily Dose Needed
Description: Magnitude was determined via a change table which provides the percentage of participants that needed a change in Daily Dose (μg/day) of -25 μg, -12.5 μg, -6.25 μg, -5.35 μg, 0 μg or +12.5 μg.
Time Frame: 2 months (± 2 weeks) after switch to sodium formulation.
Population: Participants from the intent-to-treat population, with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Levothyroxine Sodium New Formulation
Number analyzed (Participants) | 82
percentage of participants
  -25 μg change | 19.51
  -12.5 μg change | 42.68
  -6.25 μg change | 1.22
  -5.35 μg change | 1.22
  0 μg change | 32.93
  +12.5 μg change | 2.44

3. Secondary Outcome: Percentage of Participants That Obtained a Thyroid Stimulating Hormone (TSH) Between 0.4-2.5 mU/L
Description: Blood samples were collected and samples were analyzed according to the local Quality System.
Time Frame: Month 4 (± 4 weeks) after inclusion into study.
Population: Participants from the intent-to-treat population, with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Levothyroxine Sodium New Formulation
Number analyzed (Participants) | 82
percentage of participants | 57.3

4. Secondary Outcome: Absolute Serum Thyroid Stimulating Hormone Values
Description: Blood samples were collected and samples were analyzed according to the local Quality System.
Time Frame: Baseline, Month 2 (± 2 weeks) and Month 4 (± 4 weeks) after inclusion into study.
Population: Participants from the intent-to-treat population, with data available for analysis.
Measure: Mean (Inter-Quartile Range); unit: mIU/mL
Arm/Group | Levothyroxine Sodium New Formulation
Number analyzed (Participants) | 84
mIU/mL
  Baseline | 1.1 (0.59) [0.7 to 1.6]
  Month 2 (n=83) | 0.3 (1.69) [0.1 to 0.6]
  Month 4 (n=82) | 0.6 (1.09) [0.2 to 1.0]

5. Secondary Outcome: Relative Percent Change From Baseline in Serum Thyroid Stimulating Hormone
Description: Blood samples were collected and samples were analyzed according to the local Quality System. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Month 2 (± 2 weeks) and Month 4 (± 4 weeks) after inclusion into study.
Population: Participants from the intent-to-treat population, with data available for analysis.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Levothyroxine Sodium New Formulation
Number analyzed (Participants) | 83
percent change
  Month 2 | -74.5 (192.14) [-89.5 to -50.6]
  Month 4 (n=82) | -54.0 (173.36) [-75.1 to -15.5]

ADVERSE EVENTS:
Time Frame: 5 months from inclusion (all patients) or up to recovery/final status is known for AE's.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Levothyroxine Sodium New Formulation
Serious Adverse Events (participants affected / at risk) | 7/101
Other Adverse Events (participants affected / at risk) | 7/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levothyroxine Sodium New Formulation (N=101)
Cardiac failure (Cardiac disorders) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Catheterisation cardiac (Investigations) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Bladder catheterisation (Surgical and medical procedures) | 1
Hysterectomy (Surgical and medical procedures) | 1
Mastectomy (Surgical and medical procedures) | 1
Salivary gland resection (Surgical and medical procedures) | 1
Haemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levothyroxine Sodium New Formulation (N=101)
Nasopharyngitis (Infections and infestations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.